CLINICAL TRIAL: NCT04814381
Title: Evaluation of the Efficacy of a Single Infusion of Ketamine Combined With Magnesium Sulfate to Treat Refractory Chronic Cluster Headache
Brief Title: Ketamine + Magnesium for Chronic Cluster Headache (KETALGIA)
Acronym: KETALGIA
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RBHP 2020 MOISSET; 2020-003604-14 (EudraCT Number)
Record Dates: First submitted 2021-03-18; First posted 2021-03-24 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2024-10

CONDITIONS: Refractory Chronic Cluster Headache
Keywords: Chronic cluster headache; Ketamine; Magnesium
MeSH Terms: conditions — Cluster Headache | interventions — Ketamine; Magnesium Sulfate; Drug Combinations

STUDY DESIGN:
Intervention Model Description: patients will be randomised with 1:1 ratio
Who Masked: Participant, Investigator
Masking Description: infusion will be prepared by a nurse that is not blinded to the treatment and will not take part to patient evaluation. Active and control treatments are of transparent colour and will not be recognisable.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ketamine + Magnesium (Experimental): patients in the experimental group will receive 0.5mg/kg of ketamine over 2 hours, diluted in 50cc of NaCl 0.9% and 3g of magnesium sulfate over 30 minutes diluted in 250cc of NaCl 0.9%.
  Interventions: Drug: Ketamine + Magnesium sulfate (drug combination)
- Control (Active Comparator): patients in the control group will receive 25mg of hydroxyzine over 2 hours, diluted in 50cc of NaCl 0.9% and 250cc of NaCl 0.9% over 30 minutes
  Interventions: Drug: Ketamine + Magnesium sulfate (drug combination)

INTERVENTIONS:
Drug: Ketamine + Magnesium sulfate (drug combination) — A single infusion will be performed over 2 hours with 90 days follow-up.

SUMMARY:
Chronic cluster headache (CCH) is a rare primary headache disorder, defined by episodic attacks that occur for more than one year with no remission period or with remission periods lasting < 3 months (ICHD-3 criteria). In certain cases, CCH patients become drug-resistant and continue to suffer almost daily attacks.

Ketamine appears to be effective in a variety of chronic pain conditions, such as refractory headache, and can show an enhanced analgesic effect when combined with magnesium. A single infusion of ketamine-magnesium combination has been described to reduce attacks in 17 patients with rCCH. The main outcome was a comparison of the number of daily attacks two weeks prior to the infusion and one week after (days 7-8). The number of daily attacks decreased from 4.3±2.4 before treatment to 1.3±1.0 after treatment (p<0.001). 13/17 had at least 50% response. Thus, the goal of this placebo-controlled study is to try to confirm these findings.

DETAILED DESCRIPTION:
Chronic cluster headache (CCH) is a rare primary headache disorder, defined by episodic attacks that occur for more than one year with no remission period or with remission periods lasting < 3 months (ICHD-3 criteria). In certain cases, CCH patients become drug-resistant and continue to suffer almost daily attacks.

Ketamine appears to be effective in a variety of chronic pain conditions, such as refractory headache, and can show an enhanced analgesic effect when combined with magnesium. A single infusion of ketamine-magnesium combination has been described to reduce attacks in 17 patients with rCCH. The main outcome was a comparison of the number of daily attacks two weeks prior to the infusion and one week after (days 7-8). The number of daily attacks decreased from 4.3±2.4 before treatment to 1.3±1.0 after treatment (p<0.001). 13/17 had at least 50% response. Thus, the goal of this placebo-controlled study is to try to confirm these findings.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* Chronic cluster headache diagnosis made according to ICHD-3 criteria
* A mean of at least 2 attacks/day during the 14 days before infusion
* Insufficient efficacy or intolerance or contra-indication to the use of the 3 main validated treatments (verapamil, lithium and sub-occipital steroids injections)
* Stable preventive treatment for at least 7 days before infusion

Exclusion Criteria:

* Pregnant or lactating woman
* Contra-indication to ketamine use (uncontrolled high blood pressure, stoke history, severe cardiac failure)
* Ketamine use during the previous year
* Hypersensitivity to the product or their metabolites
* Severe renal insufficiency (creatinine clearance < 30ml/min)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2021-09-15 (Actual); Primary Completion 2026-09-15 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in weekly attacks between day 7 - day 13 period compared to the pre-treatment period | pre-treatment period and day 7-day 13 post-treatment period
  Evaluate the efficacy of a single infusion of ketamine combined with magnesium sulfate compared to a control group receiving hydroxyzine (active placebo) in terms of weekly attacks between day 7 and day 13 period and pre-treatment period

SECONDARY OUTCOMES:
Proportion of 30% responders | day 7 to day 90
  proportion of 30% responders at various time points according to the attack diary
Proportion of 50% responders | day 7 to day 90
  proportion of 50% responders at various time points according to the attack diary
Proportion of 75% responders | day 7 to day 90
  proportion of 75% responders at various time points according to the attack diary
week by week attacks frequency | day 0 to day 90
  Area under the curve (AUC) for daily attacks evaluated each week between D0 and D90 (attacks diary)
patient global impression of change (PGIC) | Day 15
  PGIC will be completed and compared between the 2 groups
patient global impression of change (PGIC) | Day 90
  PGIC will be completed and compared between the 2 groups
Infusion's safety | day 0
  proportion of patients in each group reporting any side effect during or in the 24 hours after infusion (together with the type and intensity of these side effects)
Infusion's safety | day 1
  proportion of patients in each group reporting any side effect during or in the 24 hours after infusion (together with the type and intensity of these side effects)
Proportion of patients necessitating rescue therapy | Day 15
  Proportion of patients necessitating rescue therapy (infusion of ketamine combined with magnesium)
Treatment response according to initial magnesemia | day 7
  magnesemia on the infusion day (D0) will be correlated with 50% response at D7-8 among patients receiving active treatment
Treatment response according to initial magnesemia | day 8
  magnesemia on the infusion day (D0) will be correlated with 50% response at D7-8 among patients receiving active treatment
Attacks treatment consumption | day 0 to day 90
  Daily attacks treatment consumption (injectable sumatriptan and oxygene)
Direct medical cost | day 0 to day 90
  Direct medical cost (treatments, consultations, hospitalisations) in each group and cost effectiveness ratio taking 50% responder rate as efficacy criteria
Anxiety evolution | Day 15
  comparison of anxiety (evaluated via the HAD scale) between groups
Anxiety evolution | Day 90
  comparison of anxiety (evaluated via the HAD scale) between groups
depression evolution | Day 15
  comparison of depression (evaluated via the HAD scale) between groups
depression evolution | Day 90
  comparison ofdepression (evaluated via the HAD scale) between groups
Change in weekly attacks between day 14 - day 20 period compared to the pre-treatment period | pre-treatment period and day 14 - day 20 post-treatment period
  Evaluate the efficacy of a single infusion of ketamine combined with magnesium sulfate compared to a control group receiving hydroxyzine (active placebo) in terms of weekly attacks between day 14 and day 20 post-reatment period and pre-treatment period. The number of weekly attacks will be evaluated using a attacks diary that patients will complete every day.
Change in weekly attacks between day 21 - day 27 period compared to the pre-treatment period | pre-treatment period and day 21 - day 27 post-treatment period
  Evaluate the efficacy of a single infusion of ketamine combined with magnesium sulfate compared to a control group receiving hydroxyzine (active placebo) in terms of weekly attacks between day 21 and day 27 post-reatment period and pre-treatment period. The number of weekly attacks will be evaluated using a attacks diary that patients will complete every day.
Change in weekly attacks between day 28 - day 34 period compared to the pre-treatment period | pre-treatment period and day 28 - day 34 post-treatment period
  Evaluate the efficacy of a single infusion of ketamine combined with magnesium sulfate compared to a control group receiving hydroxyzine (active placebo) in terms of weekly attacks between day 28 and day 34 post-treatment period and pre-treatment period. The number of weekly attacks will be evaluated using a attacks diary that patients will complete every day.
Adverse events assessment | D0 to D90
assessment of blind quality | Day 0
  A blinding questionnaire will be systematically used to assess the quality of the blind. It will be completed by each patient 30 minutes after the end of the 1st infusion at day 0 (Visit 1). The patient will be asked what treatment he thinks he has received.

CONTACTS AND LOCATIONS:
Overall Officials: Xavier MOISSET, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (14):
- France (14):
  - CH Annecy Genevois, Annecy
  - Polyclinique Jean Villar, Bruges
  - CHU de Clermont-Ferrand, Clermont-Ferrand
  - CHRU De Lille, Lille
  - Hospices civils de Lyon, Hôpital Pierre Wertheimer, Lyon
  - AP-HM Marseille, Marseille
  - Clinique Beau Soleil, Montpellier
  - CHU de Montpellier, Montpellier
  - CHU Nantes, Hopital Nord Laennec, Nantes
  - Hôpital Lariboisière, Paris
  - CHU Rouen, Rouen
  - Hopital de Hautepierre, Strasbourg
  - Hopital Pierre Paul Riquet, Toulouse
  - CHU Grenoble-Alpes, Voiron

IPD SHARING:
Plan to Share IPD: No